CLINICAL TRIAL: NCT05494138
Title: Nutriomics and Artificial Intelligence Nutrition Obesity Cohort
Status: Recruiting | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2022-0645
Record Dates: First submitted 2022-08-07; First posted 2022-08-09 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The obese group: Obese patients (BMI ≥25 kg/m2) with chronic diseases such as cardiovascular disease, hypertension, diabetes, and metabolic syndrome. More than 10% of the patients in the obese group will be patients with a BMI ≥30.
- The control group: Adults with BMI 18.5~24.9 kg/m2.

SUMMARY:
The purpose of this study is to establish a prospective cohort. From registration to the 5th year, basic investigation, specific examinations for cardiovascular and metabolic disease, basic blood tests, collection of human material samples, and clinical event follow-up are conducted yearly. The obese group will be examined yearly, and telephone follow-up will be conducted if necessary. The control group will participate in the baseline survey once enrollment and clinical event follow-up by phone will be conducted annually thereafter. From the 6th year, only clinical event follow-up will be conducted.

DETAILED DESCRIPTION:
The obese group will enroll 500 people within 1 year of study initiation and follow-up annually. The control group will enroll 30 patients a year for 5 years.

ELIGIBILITY:
Inclusion criteria for the obese group

1. Adults 19 years of age or older
2. Obese patients with chronic diseases such as cardiovascular disease, hypertension, diabetes, and metabolic syndrome (BMI ≥ 25 kg/m2, [BMI ≥ 30 kg/m2, including 10% or more])

Inclusion criteria for the control group

1. Adults 19 years of age or older
2. Those with BMI 18.5~24.9 kg/m2

Exclusion criteria for the obese group

1. Serious non-cardiovascular disease with life expectancy less than 6 months
2. Pregnant or suspected of being pregnant or are lactating
3. Patients within 3 months of organ transplantation
4. Patients currently being treated for acute transplant rejection
5. Patients treated for acute coronary syndrome (myocardial infarction, unstable angina) and discharged within 6 months
6. Patients with acute cerebral infarction within 6 months of being hospitalized and discharged
7. Type 1 Diabetes
8. Patients taking steroids, female hormones
9. Those who have difficulty using smartphones

Exclusion criteria for the control group

1. Serious non-cardiovascular disease with life expectancy less than 6 months
2. Pregnant or suspected of being pregnant or are lactating
3. Persons who are continuously taking medications prescribed by a doctor due to chronic diseases excluding hypertension and dyslipidemia
4. Within 5 years of diagnosis of malignant tumor
5. Those who have difficulty using smartphones

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The obese group will be selected from patients who visit the department of cardiology or endocrinology for the management of chronic diseases. The control group will be selected from among those who voluntarily participate in the epidemiological study of normal participants.
Sampling Method: Non-Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2041-08-31 (Estimated)

PRIMARY OUTCOMES:
Differences of nutriomics according to obesity phenotypes | At five years of study
  Cross-sectional analysis of nutriomics of normal control group and obese patients

SECONDARY OUTCOMES:
Clinical events | three years, four years, five years, etc
  A composite of all-cause mortality, cardiovascular mortality, non-fatal myocardial infarction, non-fatal stroke, revascularization of coronary artery, and heart failure hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Sungha Park, Principal Investigator — Division of Cardiology, Severance Hospital, Yonsei University College of Medicine
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
When there is a request for data sharing from other researchers, the principal investigator will review it and decide whether to share it or not.